CLINICAL TRIAL: NCT02088853
Title: Small Intestinal Adaptation to Isocaloric Diets Dominated Either by Fats or Carbohydrates
Brief Title: Diet Induced Intestinal Mucosal Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BUTTER
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy Conditions
Keywords: intestinal; metabolic control; mucosa; human; diet
MeSH Terms: interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First high fat diet, then high carbohydrate diet (Experimental): had; first sixty percent fat as the energy source, then sixty percent carbohydrates
  Interventions: Dietary Supplement: high fat diet (hfd), then high carbohydrate diet
- First, high carb diet, then high fat diet (Experimental): had; first sixty percent carbohydrates as the energy source, the sixty percent fat
  Interventions: Dietary Supplement: high carbohydrate diet, then high fat diet

INTERVENTIONS:
Dietary Supplement: high fat diet (hfd), then high carbohydrate diet — Sixty % of the energy content is based on fat, then sixty % of the energy content is based on carbohydrates
  Arms: First high fat diet, then high carbohydrate diet
Dietary Supplement: high carbohydrate diet, then high fat diet — Sixty % of the energy content is based on carbohydrates, then sixty % of the energy content is based on fat
  Arms: First, high carb diet, then high fat diet

SUMMARY:
Human beings are 'omnivores' meaning that all principal components of food (i.e. the macronutrients: carbohydrates, fat, proteins) can be assimilated by the gastrointestinal tract. When the gut mucosa is exposed to dietary changes it adjusts its functional behaviour. For example, a fatty diet demands certain digestive mechanisms, whereas others are needed to take care of a carbohydrate rich diet. Such dietary induced changes in appearance and functionality of the small intestinal mucosa have been described in animals but only little is known about it in man. The present project aims at elucidating in man if a 2 weeks diet dominated by either fat or carbohydrates, but with similar energy content, is associated with changes in the small intestinal mucosal appearance and metabolic signalling capacity.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteer not taking prescribed medications BMI ≤25 kg/m2

Exclusion Criteria:

BMI ≥26 kg/m2 smoker previous or current gastrointestinal disease significant abdominal surgery pregnancy/breast feeding drug intolerance of importance (particularly opiates and midazolam used during endoscopy) history of drug addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fändriks, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Dept of Gastrosurgical R&E, Sahlgrenska Universityhospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Elebring E, Wallenius V, Casselbrant A, Docherty NG, Roux CWL, Marschall HU, Fandriks L. A Fatty Diet Induces a Jejunal Ketogenesis Which Inhibits Local SGLT1-Based Glucose Transport via an Acetylation Mechanism-Results from a Randomized Cross-Over Study between Iso-Caloric High-Fat versus High-Carbohydrate Diets in Healthy Volunteers. Nutrients. 2022 May 7;14(9):1961. doi: 10.3390/nu14091961. PMID 35565929

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant had BMI ≥25 kg/m2 and was excluded
Groups:
- First High Fat Diet, Then High Carbo Diet: Experimental: First high fat diet, then high carbohydrate diet had; first sixty percent fat as the energy source, then sixty percent carbohydrates
- First High Carb Diet, Then High Fay Diet: Experimental: First, high carb diet, then high fat diet had; first sixty percent carbohydrates as the energy source, the sixty percent fathigh carb diet: Sixty % of the energy content is based on carbohydrates.
Period: Overall Study
Arm/Group | First High Fat Diet, Then High Carbo Diet | First High Carb Diet, Then High Fay Diet
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: * one participant showed a BMI ≥25kg/m2 and was excluded (exclusion criterion)
  * another participant became pregnant during the study (exclusion criterion)
Groups:
- All Study Participants: The subjects had 2 periods of either
  1. first a high fat diet followed by a high carbohydrate diet or
  2. first a high carbohydrate diet followed by a high fat diet
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Mucosal Surface Enlargement
Description: The enlargement of the luminal surface area is a morphometric factor, defined as the percentage of the mucosal surface (one dimension in arbitrary units) in relation to the relatively flat area of the muscular mucosae layer from the same histological cuts. Unit: % of the muscular mucosae.
Time Frame: Appearance after 2 weeks of each diet
Population: healthy volunteers
Measure: Mean (Standard Error); unit: percentage of muscular mucosae
Groups:
- High Fat Diet: had; sixty percent fat as the energy source
  high fat diet (hfd): Sixty % of the energy content is based on fat.
- High Carb Diet: had; sixty percent carbohydrates as the energy source
  high carb diet: Sixty % of the energy content is based on carbohydrates.
Arm/Group | High Fat Diet | High Carb Diet
Number analyzed (Participants) | 15 | 15
percentage of muscular mucosae | 10.2 (2.0) | 9.9 (1.9)
Statistical Analysis 1: Comparison: High Fat Diet vs High Carb Diet; Test type: Superiority — Wilcoxon test; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Glucose Induced Electrogenic Responses In-vitro
Description: Jejunal mucosal biopsies are mounted as a sheet between two different (glucose-free) physiological solutions (in so called Ussing chambers). The electrogenic response to glucose will be measured as follows: Baseline ion-transporting capacity for the luminal to serosa side will be measured as the epithelial current (Iep) in the absence of glucose (unit; µA/cm2). Addition of 10mM glucose on the luminal side increases the ion-transporting capacity. This level will be divided with preceding baseline ion-transporting capacity and is presented as % change from the baseline secretion. The sensitivity of this response to phloridzin is given to confirm to what extent the glucose transporter SGLT1 is involved. Only the completed pairs (high fat diet versus high carbohydrate diet) will be analyzed.
Time Frame: The condition after 2 weeks of each diet
Population: Four pairs of jejunal mucosae were excluded due to technical errors.
Measure: Mean (Standard Error); unit: % change from baseline
Groups:
- High Carbohydrate Diet; High Fat Diet: Mucosal biopsies are mounted in mini Ussing chambers. Ion-transporting capacity via SGLT-1 transported is reflected when switching from a glucose-free to glucose-containing luminal solution. Selectivity of transporter is confirmed by addition of phloridzin.
  Only the values from corresponding pairs (high carb diet and high fat ditet) will be included in the analysis.
Arm/Group | High Carbohydrate Diet | High Fat Diet
Number analyzed (Participants) | 11 | 11
% change from baseline | 42 (12) | 2 (13)
Statistical Analysis 1: Comparison: High Carbohydrate Diet; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Glycemic Control Following a Test Meal
Description: Blood concentrations of glucose are assessed over 2 hours following a mixed test meal.
Time Frame: The condition after 2 weeks of each diet
Measure: Mean (Standard Error); unit: mMol/L * 120 min
Groups:
- High Carbohydrate Diet: A mixed meal is given and the glycemic values are measured intravenously over 120 min.
- High Fat Diet: A mixed meal is given and the glycemic values are measured intravenously over 120 minutes.
Arm/Group | High Carbohydrate Diet | High Fat Diet
Number analyzed (Participants) | 15 | 15
mMol/L * 120 min | 699 (24) | 732 (25)
Statistical Analysis 1: Comparison: High Carbohydrate Diet vs High Fat Diet; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 8 weeks, in other words: 1w from introductory examination/randomisation, + 2w for the first diet period + 2w for habitual food choice + 2w for the first diet period + 1w for post study.
Description: Healthy, normal weight volunteers
Groups:
- All Study Participants: had sixty percent fat as the energy source during 2w, then sixty percent carbohydrates during 2w
  or
  had sixty percent carbohydrates as the energy source during 2w, then sixty percent fats during 2w
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes